CLINICAL TRIAL: NCT05241769
Title: The Influence of Inhaled CorticoSteroids Adherence on Treatment Response to Mepolizumab in Severe Eosinophilic Asthma (CSAREA Study)
Brief Title: The Influence of Inhaled CorticoSteroids Adherence on Treatment Response to Mepolizumab in Severe Eosinophilic Asthma
Acronym: CSAREA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: RRK7437
Record Dates: First submitted 2022-01-19; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Asthma; Eosinophilic
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aim is to look at the effect of the regular use of inhaled corticosteroids on the response and received from mepolizumab treatment which you are receiving or had received before.

DETAILED DESCRIPTION:
Examine the outcomes of 250 patients who have been treated with mepolizumab within BRSAS and compare the adherence to ICS in the responders and non-responder groups. If confirmed that non-adherence to ICS was related to poor response to mepolizumab, steps then will be undertaken to better monitor and enhance adherence to ICS to improve patients outcomes and response to mepolizumab treatment.

This study will rely on retrospective analysis of medically existing data within the service ,the adherence to ICS treatment will be measured using the prescription possession ratio "PPR" Data is available in the patients' GP records and forms part of the routine clinical practice of the severe asthma clinic to monitor adherence to ICS treatment.

For a significant number of patients ,such data will be already available within patient medical records held at University Hospitals Birmingham NHS Foundation Trust (UHB), however missing data is expected and in such cases GP surgeries will be contacted to obtain the PPR. Patients will be asked to agree to access to GP records as part of the informed consent process.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years of age or higher
* Patients commenced on mepolizumab within the BRSAS network
* Patients who have at least 1 mepolizumab injection and with at least 3 months follow-up data from the time of treatment initiation
* Patients must be able and willing to give informed consent to participate in the study . An Interpreter will be provided for those patients where English is not their first language.

Exclusion Criteria:

* Refusal or inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Birmingham Regional Severe Asthma
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
To assess the influence of inhaled corticosteroids (ICS) adherence on treatment response to mepolizumab in severe eosinophilic asthma | 20 months
  We will measure the adherence to inhaled corticosteroids treatment (ICS) during the period when patients were treated with the biologic treatment mepolizumab. Adherence to ICS will be measured in the form of prescription possession ratio (PPR) in which the number of prescription picked up by patients is divided by the expected number to be used in a specified period of time (one year). Adherence will be defined as a PPR of =>70%. Mepolizumab responser group will be defined as those achieving reduction in the use of maintenance oral corticosteroids (OCS) and/or frequency of severe asthma exacerbations require OCS treatment by =>50%. The adherence rates to ICS as measured by PPR in the mepolizumab responder and non-responder groups will be compared to find out if ICS non-adherence reduce response to meplizumab treatment in patients with severe eosinophilic asthma

SECONDARY OUTCOMES:
to describe baseline demographic and clinical characteristics of severe eosinophilic asthma patients treated with mepolizumab in the BRSAS network | 20 months
  General demographics and clinical characteristics of the mepolizumab treated population in BRSAS will be presented and these will include age, gender, ethnicity, asthma severity measures in the form of symptoms, lung function, treatment use and requirement for maintenance oral corticosteroids, exacerbation frequency, admissions and emergency department visits.
To describe the overall response and clinical outcomes to mepolizumab therapy in the BRSAS population. | 20 months
  Treatment response to mepolizumab will be assessed at the one year end of treamtent in which patients will be labelled as responder if they achieved a meaningful clinical response using NICE criteria of reducing severe exacerbation frequency by 50% or more and/or reducing the dose of maintenance OCS by similar magnitude. The overall response rate in the 250 patients will be reported as a responder proportion. The overall benefit from treatment in the form of its effect on asthma measures such as asthma control questionnaire, lung function, biomarkers of blood eosinophils and exhaled nitric oxide, admissions, emergency department visits and any reported side effects will be reported.
to measure the frequency of severe exacerbations requiring oral corticosteroids treatment in patients treated with mepolizumab in patients with high/low fraction exhaled nitric oxide groups. | 20 months
  Fraction exhaled nitric oxide (FeNO) is an inflammatory marker of asthma. FeNO has been used as a marker of non-adherence to inhaled corticosteroids (ICS). Patients non-adherent to ICS tend to have high FeNO as ICS often potently suppress FeNO. High FeNO level despite ICS treatment would indicate continuing active asthma airway inflammation and increased risk of exacerbation. We will divide patient groups into high and low FeNO groups using different cut-off levels of 25,35,50 parts per billion (PPB). FeNO high and low groups will be compared in terms of severe asthma exacerbation frequency to determine if persistent high FeNO is associated with exacerbations. An increase in exacerbation frequency in FeNO-high patients would indicate that FeNO can be used as surrogate marker of ICS non-adherence or inadequate suppression of T2 asthma inflammation due to ICS resistance with both may drive incomplete response to mepolizumab treatment.
To determine the response rate to mepolizumab in FeNO high and FeNO low groups (using variable cut off levels). | 20 months
  As per outcome 4 we will categorise patients as FeNO high and FeNO low groups using cut off levels of 25,35,50 ppb and compare the response to mepolizumab in the FeNO high/low groups. Response to empolizumab will be determined as described in outcome 3. Patients continue to express high FeNO despite mepolizumab treatment are likely to have the disadvantage of unsuppressed type 2 asthma inflammation and therefore are at risk of exacerbation and are probably less likely to have be responder to mepolizumab. This assertion however has not been previously definitely confirmed and this analysis will help in clarifying this matter further.
To investigate the relationship between FeNO and ICS dose in patients on mepolizumab treatment. | 20 months
  We will look at the prescribed dose of inhaled corticosteroids (ICS) and its relation to FeNO level. ICSs are potent suppressors of FeNO and it is expected therefore that patients receiving regular ICS treatment will express lower FeNO level than those not on ICS or are non-adherent to ICS. It is not certain if there is actual relation between ICS dose as measured in microgram of beclomethasone equivalent daily dose FeNO level as too many variables may affect this (for example, non-adherence to ICS, ICS resistant patient groups, variable delivery efficiency of the drug to the airways). Therefore in this analysis we will perform correlation and association analysis of mean FeNO level and mean ICS daily dose (beclomethasone equivalent) to explore the effect of ICS of FeNO in this group of patient who are also treated with mepolizumab at the same time.
To investigate the relationship between the prescription possession ratio (PPR) of inhaled corticosteroids (ICS) and FeNO level in patients on mepolizumab treatment. | 20 months
  One of the measures of treatment adherence to preventer therapy (ICS) used in clinical practice the prescription possession ratio (PPR) (=total number of ICS inhaler prescriptions picked up in the 12 months period whilst on mepolizumab / expted number to be picked up in this period). A PPR ratio of 70% or higher has been used in literature to indicate adequate adherence and thefore this cut-off level has been accepted in current clinical practice in UK (NHSE severe asthma tool kit). Complementing the analysis of relationship between mean ICS dose and mean FeNO (outcome 6), the analysis of PPR relation with FeNO is expected to be more accurate as it does take into consideration the potential strong confounder of ICS non-adherence. If confirmed that PPR is related to FeNO level then interventions to enhance adherence to ICS can be instituted to suppress FeNO and in turn improve asthma outcomes.
To determine the mepolizumab response rate in the ICS adherent versus non-adherent patients (at 70% ICS PPR cut off level). | 20 months
  Response rate to mepolizumab as measured by effective reduction in either maintenance oral corticosteroids dose (OCS) and /or frequency of OCS requiring exacerbations at the one year end of mepolizumab treamtent, will be compared in patients who are adherent to ICS (adherent = those who has precription possession ratio (PPR) of 70% or higher) or non-adherent. The hypothesis here is that ICS non-adherence can influence response rate to mepolizumab as part of the asthma inflammation no suppressed enough by mepolizumab will persist due to lack of adequate ICS treatment and therefore mepolizumab will less likely work in patients not taking ICS adequately. If this is demonstrated through this analysis, again more emphasis will be put to enhance the adherence to ICS that would then improve response rate to mepolizumab.
To compare mean inhaled corticosteroids (ICS) daily dose and prescription possession ratio (PPR) in the period before and on mepolizumab treatment. | 20 months
  In this analysis we will compare the mean ICS daily dose and PPR in the 12 months before and the 12 months on mepolizumab treatment. Several studies showed that initiation of biologic treatment such as mepolizumab can result in reduced adherence to ICS. Asthma improvement due to mepolizumab with reduced daily symptoms of asthma may result in patients not persevering with their daily regular ICS treament or patient may feel that a potent asthma injection such as mepolizumab is sufficient and do not need ICS (often despite medical advice). In this analysis we will therefore explore if there is evidenc of change in behaviour in terms of PPR before and on biologic treamtent period and if demonstrated then factors driving such change in adherence will require further exploration.
To explore patient characteristics and predictors of poor ICS adherence | 20 months
  We will compare clinical characteristics of patients with poor ICS adherence (as measured by those with PPR ration of <70%) to the adherent groups with aim to identify an predictors of non-adherence that may prompt further research into drivers of non-adherence to eventually develop tools and intervention to address these to improve patients outcomes. Clinical charactersitics that would include age, gender, ethnicity, asthma symptoms control level, quality of life, exacerbatin frequency, use of maintenance OCS, lung function and others will be explored in this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Adel Mansur, Study Director — UHB

IPD SHARING:
Plan to Share IPD: No